CLINICAL TRIAL: NCT01986660
Title: Open-Label, Maximum-Dose Pharmacokinetic Study of 7.5% Ibuprofen Cream (SST-0225) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Strategic Science & Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: SST0225-US-011-001
Record Dates: First submitted 2013-10-29; First posted 2013-11-18 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2014-01

CONDITIONS: Healthy
Keywords: Pharmacokinetic Study

ARMS (1):
- Ibuprofen Cream (SST-0225) (Experimental)
  Interventions: Drug: Ibuprofen Cream (SST-0225)

INTERVENTIONS:
Drug: Ibuprofen Cream (SST-0225)

SUMMARY:
The purpose of this study is to evaluate how Ibuprofen Cream (SST-0225) is absorbed and eliminated by the body under defined maximum dosing conditions and to evaluate the safety under these conditions.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent form
* Men, women, 18 to 55 years
* Females must not be pregnant or plan to become pregnant
* BMI 18 to 30 kg/m2
* Past or non-smoker
* High probability of compliance with completion of study
* Healthy as determined by investigator based on medical history, physical exam, clinical laboratory tests, vital sign measurements, ECGs

Exclusion Criteria:

* Presence or history of disorder that could interfere with completion of study
* Unstable medical condition
* Surgical or medical condition that may interfere with absorption, distribution, metabolism or excretion of test drug
* Positive Hep B, Hep C and/or HIV test
* Positive urine drug screen
* Any history of skin disorders, including psoriasis, eczema, tattoos, significant scarring, healing wounds, skin lesions on knees or elbows
* Significant disease
* Any clinically important deviation from normal limits in physical exam, vital sign measurements, 12 lead ECG, clinical laboratory test
* History of drug abuse with 1 year
* History of alcoholism with 1 year
* Use of prescription medications or ibuprofen within 30 days of Day 1, use of OTC drugs, herbal supplements and vitamins within 14 days of Day 1.
* Use of investigational drug within 30 day of Day 1
* Acute disease state within 7 days of Day 1
* Consumption of grapefruit or grapefruit containing products within 72 hours of Day 1
* Tobacco use/caffeine use within 48 hours of Day 1

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Cmax, Tmax, Trough Concentrations Days 2 to 8, AUC 0-24, Steady State, T1/2 | 9 days

SECONDARY OUTCOMES:
Clinical laboratory change from baseline | 14 days
Modified Berger Bowman Skin Assessment | 14 days
Vital Signs | 14 days
Adverse Events | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- SST Investigational Site, New York, New York, United States